CLINICAL TRIAL: NCT03807570
Title: A 12 Weeks, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety Morus Alba L. Extract on Improvement of Blood Flow
Brief Title: Efficacy and Safety Morus Alba L. Extract on Improvement of Blood Flow
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BA-BF-MBE
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Blood Flow
Keywords: Morus Alba L. Extract; Clinical Trial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morus Alba L. extract (Experimental): Morus Alba L. extract 30 ml/day for 12 weeks
  Interventions: Dietary Supplement: Morus Alba L. Extract
- Placebo (Placebo Comparator): Placebo 30 ml/day for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Morus Alba L. Extract — Morus Alba L. Extract 30 ml/day for 12 weeks.
  Arms: Morus Alba L. extract
Dietary Supplement: Placebo — Placebo 30 ml/day for 12 weeks.
  Arms: Placebo

SUMMARY:
The effect of 12 weeks intake of Morus alba L. on blood circulation improvement and related indicators is assessed compared to placebo intake.

DETAILED DESCRIPTION:
This study was a 12 weeks, randomized, double-blind, placebo-controlled human trial. Hundred subjects were randomly divided into Morus alba L. extract or a placebo group. Blood was collected and changes in blood circulation related indicators were observed.

ELIGIBILITY:
Inclusion Criteria:

* Those with a fasting total cholesterol of 200~239 mg/dL
* Those with a fasting LDL-cholesterol of 130~159 mg/dL
* Those with a fasting blood sugar of 100~125 mg/dL
* Those with a SBP of 120~139 mmHg
* Those with a BMI of 25~29.9 kg/m^2
* Waist Hip Ratio (WHR) is 0.9 or more for males and 0.85 or more for females

Exclusion Criteria:

* Those with platelet aggregation and significant disability

  * The platelet count is less than 100,000/μL or more than 500,000/μL
  * The Hematocrit is less than 25%
* BMI is less than 18.5kg/m^2 or greater than 30kg/m^2
* Those with clinically significant severe cardiovascular, endocrine, immune, respiratory, liver, biliary, renal and urinary tract, neuropsychiatry, musculoskeletal, inflammatory and hematologic and gastrointestinal disorders
* Those with a history of clinically significant hypersensitivity to mulberry
* Those who have been taking platelet function, blood circulation improvement and hyperlipidemia related medicines, health functional food or herbal medicine continuously for more than 7 days within one month before screening
* Those who have received antipsychotic medication within 2 months before screening
* Those who participated in other clinical trials within 3 months before screening
* Women receiving hormone replacement therapy
* Laboratory test by show the following results

  * AST, ALT > Reference range 3 times upper limit
  * Serum Creatinine > 2.0 mg/dL
* Pregnancy or breast feeding
* Those who doesn't accept the implementation of appropriate contraception of a childbearing woman
* Principal Investigator judged inappropriate for participation in study because of Laboratory test result, etc.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-12 (Actual); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
Changes of Reactive Hyperemia Index | 12 weeks
  Reactive Hyperemia Index was measured in study visit 1(0 week) and visit 3(12 weeks).
Changes of Platelet function assay | 12 weeks
  The whole blood with anticoagulant (sodium citrate) is passed through the capillary and the membrane to assess the degree of platelet adhesion to this membrane and the degree of occlusion of the capillary.

SECONDARY OUTCOMES:
Changes of blood flow indices: PAI-1, t-PA | 12 weeks
  Blood flow indices(PAI-1, t-PA) were measured in study visit 1(0 week) and visit 3(12 weeks).
Changes of Pulse wave | 12 weeks
  Measured using a pulse wave measuring device (uBioClipTM; BiosenseCreative Co., Ltd., Seoul, Korea) and measured three times, the average value of the measured values is indicated.
Changes of Oxidation stress index: Oxidized LDL | 12 weeks
  Oxidation stress indices(Oxidized LDL) was measured in study visit 1(0 week) and visit 3(12 weeks).
Changes of Lipid peroxidation index: MDA (Malondialdehyde) | 12 weeks
  Lipid peroxidation index{MDA(Malondialdehyde)} was measured in study visit 1(0 week) and visit 3(12 weeks).
Changes of Lipid metabolism indices: Total cholesterol, Triglyceride, LDL-C, HDL-C | 12 weeks
  Lipid metabolism indices(Total cholesterol, Triglyceride, LDL-C, HDL-C) were measured in study screening and visit 3(12 weeks).
Changes of Arteriosclerosis indices: Total cholesterol/HDL-C, LDL-C/HDL-C, Triglyceride/HDL-C, (Total cholesterol-HDL-C)/HDL-C | 12 weeks
  It is calculated by the calculation formula using the lipid metabolism indicator test item.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea